CLINICAL TRIAL: NCT00445107
Title: An Open Label, Observational Study to Assess The Efficacy, Safety and Tolerability of Added Singulair in Persistent Asthma Patients With or Without Allergic Rhinitis and Long Acting B-Agonist
Brief Title: SINGULAIR (R) as Complementary Therapy to Fixed Association Regimen (0476-363)
Acronym: STAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0476-363; 2007_002
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Duration of Therapy

INTERVENTIONS:
Drug: MK0476, montelukast sodium / Duration of Treatment: 8 Weeks

SUMMARY:
The purpose of this study is to assess the treatment effect of montelukast 10mg on the primary endpoint of Asthma Control Questionnaire(ACQ), over a 8-week period, in persistent asthma patients with or without allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Patient is currently a nonsmoker and has been a nonsmoker for at least 1 year
* Patient with clinical evidence of mild/moderate asthma with or without allergic rhinitis

Exclusion Criteria:

* Patient has been treated in an emergency room for asthma within 4 weeks or has been hospitalized for asthma within 3 months prior to visit 1
* Patient with severe asthma, upper respiratory infection, sinusitis, infectious rhinitis, non-allergic rhinitis
* Patient has any active, acute, or chronic pulmonary disorder that is documented by history, physical examination

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2005-11-01 (Actual); Primary Completion 2006-05-01 (Actual); Study Completion 2006-05-17 (Actual)

PRIMARY OUTCOMES:
Change of the asthma control questionnaire scores taken over 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC